CLINICAL TRIAL: NCT01669967
Title: The Role of Intravenous (IV) Lidocaine in the Management of Chronic Neuropathic Pain of Peripheral Nerve Origin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: R11-132; 17806 (Other: University of Western Ontario)
Record Dates: First submitted 2012-06-22; First posted 2012-08-21 (Estimated); Last update posted 2019-03-15 (Actual); Status verified 2019-03

CONDITIONS: Neuropathic Pain
MeSH Terms: conditions — Neuralgia | interventions — Lidocaine; Diphenhydramine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diphenhydramine(Benadryl) (Placebo Comparator)
  Interventions: Drug: Diphenhydramine
- Lidocaine (Active Comparator)
  Interventions: Drug: Lidocaine

INTERVENTIONS:
Drug: Lidocaine — Lidocaine 5 mg/kg in 250 ml of normal saline infused over 45 minutes.
  Other Names: Xylocaine
  Arms: Lidocaine
Drug: Diphenhydramine — Diphenhydramine 50 mg in 250 ml of normal saline infused over 45 minutes.
  Other Names: Benadryl
  Arms: Diphenhydramine(Benadryl)

SUMMARY:
Pain as a result of nerve injury (neuropathic pain) is a particularly severe form of chronic pain. Common examples of neuropathic pain are pain due to diabetes and shingles. There is good evidence that an intravenous infusion of lidocaine (local anesthetic) is useful for the management of neuropathic pain in the short term - up to six hours.

DETAILED DESCRIPTION:
This study will examine the role of intravenous lidocaine in the relief of neuropathic pain over four weeks following infusion compared to an active placebo infusion of diphenhydramine(Benadryl) in normal saline. If we can show that intravenous lidocaine provides sustained benefit for up to one month, this will be a major advance in the management of individuals suffering from neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic neuropathic pain due to diabetes mellitus or herpes zoster and a score of 4/10 or greater on the DN4 questionnaire.
* Moderate to severe pain as defined by screening average pain intensity of 5 or greater on a 0-10 numerical rating scale.
* Neuropathic pain duration of at least 6 months.

Exclusion Criteria:

* Presence of clinically significant cardiac disease.
* Poorly controlled seizure disorder.
* Significant psychiatric disorder.
* History of allergy to lidocaine or any other amide local anesthetic
* History of allergy to diphenhydramine.
* Prior treatment with a local anesthetic infusion.
* Neuropathic pain due to cancer or complex regional pain syndrome
* Language barrier or cognitive impairment that would preclude understanding of the study and filling out of questionnaires
* Lack of a driver to transport the patient to and from the pain clinic.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline Pain scores on the Visual Analog Scale at 4 weeks | every 24 hours for four weeks post-infusion

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale | obtained baseline, 24 and 72 hours and then weeks 1,2,3, and 4
Modified Brief Pain Inventory | obtained baseline, 24, 72 hours and then weeks 1,2,3 and 4
Leeds Sleep Evaluation Questionnaire | obtained baseline, 24, 72 hours and then weeks 1,2,3 and 4
Patient Global Satisfaction with Treatment and Impression of Change | obtained baseline, 24, 72 hours and then weeks 1,2,3 and 4
Side Effects | obtained baseline, 24, 72 hours and then weeks 1,2,3 and 4
Quality of Life Health Outcome Instrument | obtained baseline, 24, 72 hours and then weeks 1,2,3 and 4

CONTACTS AND LOCATIONS:
Overall Officials: Dwight Moulin, Dr., Principal Investigator — University of Western Ontario, Canada
Locations (1):
- St. Joseph's Health Care, London, Ontario, Canada

REFERENCES:
- [Derived] Moulin DE, Morley-Forster PK, Pirani Z, Rohfritsch C, Stitt L. Intravenous lidocaine in the management of chronic peripheral neuropathic pain: a randomized-controlled trial. Can J Anaesth. 2019 Jul;66(7):820-827. doi: 10.1007/s12630-019-01395-8. Epub 2019 May 16. PMID 31098961